CLINICAL TRIAL: NCT05806073
Title: Elective vs Therapeutic Neck Dissection in Treatment of Patients With Clinical T1/2N1M0 Oral Squamous Cell Carcinoma
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SH9H-2022-T349-2
Record Dates: First submitted 2023-02-21; First posted 2023-04-10 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-03

CONDITIONS: Oral Squamous Cell Carcinoma; Neck Dissection
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Elective neck dissection (Experimental): patient underwent elective neck dissection(level I-III) as initial treatment, along with the excision of the primary tumor
  Interventions: Procedure: Elective neck dissection
- Therapeutic neck dissection (Experimental): Patient underwent therapeutic neck dissection(level I-V) as initial treatment, along with the excision of the primary tumor
  Interventions: Procedure: Therapeutic neck dissection

INTERVENTIONS:
Procedure: Elective neck dissection — patient underwent elective neck dissection(level I-III) as initial treatment, along with the excision of the primary tumor
  Arms: Elective neck dissection
Procedure: Therapeutic neck dissection — patient underwent Therapeutic neck dissection(level I-V) as initial treatment, along with the excision of the primary tumor
  Arms: Therapeutic neck dissection

SUMMARY:
Cervical lymph node metastasis is the most important prognostic factor of oral squamous cell carcinoma (OSCC). Therapeutic neck dissection (I-V region) has always been regarded as the standard scheme of neck surgery for patients with cN+ OSCC and however, it has brought obvious side effects, which seriously affects the postoperative quality of life of patients. In addition, excessive neck lymph node dissection will also affect the local immune function of patients to some extent and reduce the body's response to immunotherapy. Lymph node metastasis of primary oral squamous cell carcinoma follows certain rules. Most of the metastatic areas are I-II, and low-level metastasis is very rare. Therefore, more than 90% of patients with cN+ oral squamous cell carcinoma who have undergone Therapeutic neck dissection may have suffered from "excessive dissection of area of IV and V".

Both the long-term clinical experience of surgeons and a large number of recent retrospective studies show that elective neck dissection (I-III region) is safe enough for patients with oral squamous cell carcinoma of cN1 and part of cN2.There is clearly a need therefore for a large randomized trial that will resolve the issue either way once and for all.

DETAILED DESCRIPTION:
There are controversies on the benefits of therapeutic neck dissection (I-V region) for clinically T1-2N1M0 oral squamous cell carcinoma(cT1-2N1M0). The aim of this study is to determine the need for a randomized controlled trial in order to evaluate the safety of elective neck dissection (I-III region) for patients of cT1-2N1M0. We initiate this study, expecting 188 primary oral cancer patients to be enrolled. And we are going to randomly divide these patients into two groups: "elective neck dissection (END)" and "therapeutic neck dissection (TND)". The END group will undergo one stage surgery of END and primary tumor excision, and the TND group will be treated with one stage surgery of TND and primary tumor excision. All patients will be followed up with at least 2 years after initial treatment, and the neck recurrence rate (primary outcome measures), postoperative complication rate, quality of life and survival between groups will be compared.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven T1 or T2 N1 M0( AJCC 8th) squamous call carcinoma of tongue(except base of the tongue ), buccal mucosa, upper and lower gums, hard palate and floor of mouth;
2. No history of chemotherapy, radiotherapy or targeted therapy,for any reason before
3. No history of a prior malignancy in head and neck region
4. No history of a prior malignancy outside head and neck region in the preceding 5 years
5. Eastern Cooperative Oncology Group Performance score (ECOG PS) is 0 or 1;
6. Participants will be reliable for follow-up
7. Understanding the protocol and is able to give informed consent

Exclusion Criteria:

1. failed to obtain the signed written informed consent;
2. definite distant metastasis or other malignant tumor;
3. Previous surgical operations for primary tumors or lymph nodes in the head and neck (except biopsy);
4. previously received radiotherapy for primary tumors or lymph nodes;
5. previously received anti-tumor biological targeted therapy;
6. Chemotherapy or immunotherapy has been applied to the primary tumor in the past;
7. Patients with any malignant tumor in the past 5 years (except the cured basal cell carcinoma of the skin or cervical carcinoma in situ)；
8. Any unstable systemic disease (including active infection, uncontrolled hypertension, unstable angina pectoris, angina pectoris that started in the last 3 months, congestive heart failure, myocardial infarction that occurred in the first 12 months, serious arrhythmia requiring medical treatment, liver, kidney or metabolic diseases);
9. known human immunodeficiency virus (HIV) infection;
10. chronic diseases requiring immune preparations or hormone treatment;
11. pregnant or lactating women;
12. drug/alcohol abuse, or suffering from psychological or mental diseases that may interfere with research compliance;
13. Epilepsy patients who need medical treatment (such as steroids or antiepileptic drugs);
14. participated in other clinical trials in the past 30 days;
15. cases that the researcher thinks are not suitable for joining the group.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Estimated)
Dates: Start 2023-04 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Recurrence rate of neck | up to 2 year
  From date of randomization until the date of metastasis of ipsilateral or contralateral cervical lymph nodes

SECONDARY OUTCOMES:
Overall survival | up to 2 year
  From date of randomization until the date of death from any cause

IPD SHARING:
Plan to Share IPD: Undecided